CLINICAL TRIAL: NCT06985173
Title: Patient Satisfaction and Occlusal Adjustments in Occlusal Splints Fabricated Using Fully Digital Versus Conventional Workflow in TMD Patients. (Randomized Controlled Clinical Trial)
Brief Title: Patient Satisfaction in Occlusal Splints Fabricated Using Fully Digital Versus Conventional Workflow
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Abdelhadi, Teacher assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROSR 3-3-32025
Record Dates: First submitted 2025-05-06; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: The intervention involves the fabrication of 3D printed occlusal splint with fully digitalization technique by the aid of Jaw Tracing Device (Zebis JMA, Germany). The acquisition and scanning of the patients are done by using an intra oral scanner (Medit i700, South Korea) and designing them using a designing software (Exocad, USA). This device will be printed with a 3D printer (Anycubic) utilizing printable resin material.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal splints manufactured with Conventional workflow (Active Comparator): For the comparator group, maxillary and mandibular impressions will be made with alginate impression material, models will be poured with gypsum, facebow (Bio-art) record and interocclusal registrations will be recorded at centric by using bite registration material after patient deprogramming with Lucia jig. The models will be mounted in a semi-adjustable articulator, wax pattern fabrication on surveyed and mounted casts to be invested finally to form a clear, heated-cured acrylic resin splint
  Interventions: Device: Occlusal splints manufactured with Conventional workflow
- Occlusal splints manufactured with fully digital workflow (Experimental): The intervention involves the fabrication of 3D printing of occlusal splint with fully digitalization technique by the aid of Jaw Tracing Device (Zebis JMA, Germany). The acquisition and scanning of the patients are done by using an intra oral scanner (Medit i700, South Korea) and designing them using a designing software (Exocad, USA). This device will be printed with a 3D printer (Anycubic) utilizing printable resin material
  Interventions: Device: Occlusal splints manufactured with fully digital workflow.

INTERVENTIONS:
Device: Occlusal splints manufactured with fully digital workflow. — The intervention involves the fabrication of 3D printed occlusal splint with fully digitalization technique by the aid of Jaw Tracing Device. The acquisition and scanning of the patients are done by using an intra oral scanner and designing them using a designing software. This device will be printed with a 3D printer utilizing printable resin material
  Arms: Occlusal splints manufactured with fully digital workflow
Device: Occlusal splints manufactured with Conventional workflow — For the comparator group, maxillary and mandibular impressions will be made with Cavex CA37 alginate impression material (Cavex Holland B.V, Holland), models will be poured with gypsum (Kimberlit, Type IV Dental Stone, Protechno Spain), facebow (Bio-art) record and interocclusal registrations will be recorded at centric by using bite registration material after patient deprogramming with Lucia jig. The models will be mounted in a semi-adjustable articulator (Bio-art, A7Plus, Brazil), wax pattern fabrication on surveyed and mounted casts to be invested finally to form a clear, heated-cured acrylic resin splint
  Arms: Occlusal splints manufactured with Conventional workflow

SUMMARY:
According to published literatures, the prevalence of TMD is approximately 10% in patients over 18 years of age with a considerable proportion being women of reproductive age. The treatment of TMD presents the following goals: decreasing joint and masticatory muscle pain, increasing the range of motion in the mandible, preventing degenerative changes in the articulating tissues. Management of TMD can be either conservative or surgical treatments, the conservative treatments include analgesia, medications, physical therapy, occlusal adjustment, splint therapy, localized steam application, and external muscle massage. The occlusal splint therapy is considered a common treatment option for TMD management. Flat stabilization splint is the preferred splint for such cases. It is designed to promote occlusal stability and decrease muscles tension by altering occlusion and allowing complete seating of the condyle in centric relation.

The evolution of digital technology created new era of dentistry that successfully digitalized the traditional workflow of occlusal splints including designing and manufacturing. Furthermore, virtual facebow and dynamic jaw relation record using jaw tracking device are another digital reward. The digital workflow can offer more predictable approach for occlusal splint construction, It could eliminate the traditional technical errors and enhance the occlusal accuracy

DETAILED DESCRIPTION:
The traditional workflow of occlusal splints includes, primary impression for both arches, pouring casts, patient deprogramming and centric jaw relation record followed by mounting. Then the occlusal splint is made out of a resin that includes wax pattern fabrication on surveyed and mounted casts to be invested finally to form a clear, heated-cured acrylic resin splint. After that, it is trimmed, polished, and seated back on the duplicate of the invested casts. It is a complicated process and time- consuming constructed followed by occlusal adjustments on the articulator. That traditional approach is time consuming and prone to many technical errors. Such errors are reflected in occlusal discrepancies that are considered critical for the effectiveness of occlusal splint therapy.

Recent advancements in the field of intra-oral scanning (IOS), jaw tracking device for digitally recording the maxillomandibular relationship, maximum intercuspation, centric occlusion and the patient's mandibular motion. This technique incorporates the mandibular motion into the 3-dimensional (3D) virtual patient representation to integrate the 3D dynamic virtual patient visualization and computer-aided design/computer-aided manufacturing (CAD/CAM) may have the potential to compensate for some of the shortcomings of conventional splint therapy and deliver improved clinical results, while simplifying the workflow. Several studies have shown the improved quality and material properties of CAD/CAM splints in comparison to conventional ones, but little of them reported fully digital workflow starting from scanning of maxillary and mandibular teeth, using jaw tracking device to obtain personalized condylar motion parameters and individualized maxillary position to better simulate the actual movement of the patient in the laboratory (Revilla, Marta etal,2022) and Computer-aided design/computer-aided manufacturing (CAD/CAM) in final production of occlusal splints all of these fully digital steps may be possibly reducing the adjustment time for occlusal devices and achieving predictable efficacy.

This study aims to compare the difference, if present in patient satisfaction and the amount of occlusal adjustments in occlusal splints fabricated using fully digital versus conventional workflow.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* Complete dentition.
* Normal jaw opening.
* Intact teeth.
* No ongoing dental therapy, such as orthodontic or prosthodontic treatment.
* TMD patients with more than one of following symptoms or signs: myofascial pain and /or pain in the TMJ, myofascial pain and/or pain in the TMJ on palpation, muscles tenderness, headache or earache.
* Patients who had unsuccessfully undergone splint therapy or other TMD treatments in the past were not excluded.

Exclusion Criteria:

* Patients with systemic diseases which could affect TMJ, e.g., rheumatoid arthritis, osteoarthrosis, osteoporosis, and patients taking analgesic, muscle relaxant, or anti inflammatory drugs were excluded because such drugs could influence the results.
* Temporomandibular joint lesions found on clinical palpation or medical imaging examination.
* Jaw opening less than 3 fingers.
* Patients with occlusal dysfunctions.
* Patients with severe or moderate periodontitis.
* Unable to undergo examination or treatment due to the presence of a psychological or mental disorder.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | '' Up to 12 weeks''
  Primary outcome: patient satisfaction will be recorded using Numeric scales (TMD/NS, 10 cm), this questionnaire includes the following aspects; headaches, face pain, jaw joint pain, jaw joint noises, mastication pain, neck pain, face tension, limitation of mouth opening, complaints during mastication, and teeth sensitivity at baseline and then after 1 and 3 months. The questioner was translated into Arabic language to be understood by the patients.

SECONDARY OUTCOMES:
Amount of occlusal adjustments | Base line or day 1
  Secondary outcome: amount occlusal adjustments (representing 3-dimensional volumetric changes). After finishing of occlusal device, it will be scanned with the scanner (pre-adjustment scan). The scanning will be repeated after adjustment of the occlusal device by the clinician (post-adjustment scan). The STL files of both the pre and post adjustments scans for each occlusal device will be imported to Medit link and the two scans will be superimposed by the "best fit alignment" and "3D compare" functions will be carried out to measure the amount of intraoral occlusal adjustments (in mm) that was performed

IPD SHARING:
Plan to Share IPD: No
I am not going to share the IPD for privacy and security of the information.